CLINICAL TRIAL: NCT03359642
Title: Characterization of the Intestinal Microbiota in Patients With Inflammatory Bowel Disease and/or Spondyloarthritis and Study of the Impact of an Anti-TNF Alpha Therapy
Acronym: MIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2017/28
Record Dates: First submitted 2017-11-10; First posted 2017-12-02 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Spondyloarthritis; Crohn Disease; Ulcerative Colitis
Keywords: Microbiota; inflammatory bowel disease; inflammation; anti-TNF alpha
MeSH Terms: conditions — Spondylarthritis; Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases; Inflammation | interventions — Blood Specimen Collection; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with anti-TNF alpha (Experimental): 12 spondyloarthritis and 24 inflammatory bowel diseases patients (12 Crohn's disease and 12 ulcerative colitis), in which a first anti-TNF alpha treatment is indicated.
  Interventions: Other: blood sample; Other: stool samples; Other: food questionnaire; Other: colonoscopy; Other: VOCs profile
- mirror group (Active Comparator): A mirror group of 12 spondyloarthritis and 24 inflammatory bowel diseases patients (12 Crohn's disease and 12 ulcerative colitis), in which an "all but anti-TNF alpha or biotherapy" treatment is indicated will be included to distinguish the specific effects on microbiota of anti-TNF alpha.
  Interventions: Other: blood sample; Other: stool samples; Other: food questionnaire; Other: colonoscopy; Other: VOCs profile

INTERVENTIONS:
Other: blood sample — 14 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation
Other: stool samples — Study of the fecal microbiota
Other: food questionnaire — food questionnaire on the seven days before the collection
Other: colonoscopy — Only for patients with ulcerative colitis (in routine care)
Other: VOCs profile — Volatile Organic Compounds (VOCs) profile obtained by mass spectrometry

SUMMARY:
Spondyloarthritis and inflammatory bowel diseases are common diseases, frequently met together in overlap syndromes. Their physiopathology remains puzzling. A strong role of gut microbiota has been recently put forward to explain the development of inflammatory bowel diseases, and is suspected to play an important role in rheumatoid diseases. Anti-Tumor Necrosis Factor (anti-TNF) alpha are effective and safe drugs in the treatment of both digestive and rheumatoid inflammatory diseases. The way they work is unclear, and the clinical response to this treatment is variable. A better understanding of the pathophysiology of inflammatory bowel diseases and of the action of anti-TNF alpha is essential to an optimized care.

Our hypothesis is that the efficacy of anti-TNF alpha in spondyloarthritis and in inflammatory bowel diseases is at least partly due to its restoring action of homeostasis at the interface between gastrointestinal mucosa and intestinal microbiota, either by primary action on the digestive epithelium, allowing it to regain its control and tolerance functions toward mucosal microbiota, either by direct action on the intestinal microbiota, via an inter-reigns regulation.

The main objective of our study is to assess quantitative and qualitative changes in fecal microbiota before (D0) and 3 months after initiation of anti-TNF alpha.

DETAILED DESCRIPTION:
The investigators propose to conduct an exploratory study, on 10 spondyloarthritis and 20 inflammatory bowel diseases patients (10 Crohn's disease and 10 ulcerative colitis (UC), in which a first anti-TNF alpha treatment is indicated. At D0 and M3, intestinal microbiota will be studied by DNA16S sequencing and qPCR, via a stool sampling. Volatile Organic Compounds (VOCs) profile will be obtained by mass spectrometry. Blood lymphocytes profile will be obtained by flux cytometry. In addition, a colonoscopy will be performed at D0 for UC patients, with an endoscopic and histological assessment. A second short colonoscopy will be performed for UC patients at M3. At each time, clinical assessment will be performed.

A mirror group of 10 spondyloarthritis and 20 inflammatory bowel diseases patients (10 Crohn's disease and 10 ulcerative colitis), in which an "all but anti-TNF alpha or biotherapy" treatment is indicated will be included to distinguish the specific effects on microbiota of anti-TNF alpha.

12 patients by group will be included at M0 by anticipating that some patients will stop their treatment between M0 and M3, and consequently will be excluded from M3 sampling and from final analysis. Final analysis will be performed on 10 patients by group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Patients with the following conditions :

  * Ulcerative colitis (UC) fulfilling the ECCO criteria
  * Crohn's disease (CD) fulfilling the ECCO criteria
  * Axial or peripheral spondyloarthritis (SpA) fulfilling the Assessment of SpondyloArthritis (ASAS) criteria
* Patients naïve to anti-TNF alpha, justifying the initiation of an anti-TNF alpha treatment according to current guidelines (ECCO Inflammatory bowel disease (IBD) recommendations, the recommendations of the French Society of Rheumatology for SpA)
* Patients agreeing to sign the informed consent

Exclusion Criteria:

* Patient with an inflammatory disease other than UC, CD or SpA
* History of bowel resection or digestive stoma
* Taking antibiotics in the three months preceding the stool collection
* Patients with contraindication to treatment
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline fecal microbiota profile by DNA 16S sequencing at 3 months | At 3 months from baseline

SECONDARY OUTCOMES:
Clinical response for Crohn Disease | At baseline (day 0) and at 3 months from baseline
  Harvey-Bradshaw score
Clinical response for ulcerative colitis (UC) | At baseline (day 0) and at 3 months from baseline
  Mayo score
Clinical response for spondyloarthritis (SpA) | At baseline (day 0) and at 3 months from baseline
  BASDAI or Ankylosing Spondylarthritis Disease Activity Score (ASDAS) score
Ratio of circulating Th17 / Treg lymphocytes | At baseline (day 0) and at 3 months from baseline
Only for UC group : Analysis of endoscopic activity | At baseline (day 0) and at 3 months from baseline
  Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score
Only for UC group : Analysis of histological activity | At baseline (day 0) and at 3 months from baseline
  Riley score
Change from Baseline Volatile Organic Compounds (VOCs) profile at 3 months | At baseline (day 0) and at 3 months from baseline
  VOCs levels will be obtained from exhaled air samples analyzed by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BAZIN, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Rodolphe THIEBAUT, Prof, Study Chair — University Hospital, Bordeaux; Pauline RIVIERE, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service d'Hépato-gastroentérologie, Pessac, France